CLINICAL TRIAL: NCT00904098
Title: Effectiveness And Safety Of Frovatriptan For The Management (Acute Treatment)Of Menstrual Migraine
Brief Title: Effectiveness And Safety Of Frovatriptan For The Management (Acute Treatment) Of Menstrual Migraine
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Endo Pharmaceuticals (Industry)
Responsible Party: Sr. Director, Clinical R&D, Endo Pharmaceuticals Inc.
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EN3266-401
Record Dates: First submitted 2009-05-15; First posted 2009-05-19 (Estimated); Last update posted 2010-02-15 (Estimated); Status verified 2010-02

CONDITIONS: Menstrual Migraine (MM) Headaches
Keywords: migraine
MeSH Terms: conditions — Headache; Migraine Disorders | interventions — frovatriptan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Frovatriptan (Experimental): Frovatriptan 2.5 mg oral tablet
  Interventions: Drug: Frovatriptan
- Usual Care (Active Comparator): Usual care includes the current treatment used to treat all episodes of migraine headache
  Interventions: Drug: Usual Care

INTERVENTIONS:
Drug: Frovatriptan — This study employed a prospective, non-randomized, open-label single-sequence design. The study was conducted in two phases:
  1. A Usual Care phase (approximately 1 month in duration) included one menstrual period during which female patients treated all episodes of migraine headaches using their current treatment (referred to as the Baseline phase in the protocol)
  2. An Acute Treatment phase (approximately 1 month in duration), following the Usual Care phase, included one menstrual period during which female patients used frovatriptan 2.5 mg to treat all episodes of migraine headache when their headache reached IHS Grade 1. If needed, a second dose of frovatriptan 2.5 mg was administered; however, this second dose could not be administered within 2 hours of the initial dose (i.e., there must have been at least 2 hours between doses of frovatriptan). The total daily dose of frovatriptan was not to exceed 3 tablets over a 24-hour period.
  Arms: Frovatriptan
Drug: Usual Care — Current treatment used to treat all migraine headaches
  Arms: Usual Care

SUMMARY:
Females 18 years of age or older with at least one year history of menstrual migraine (MM) headaches participated in a Phase 4 clinical trial to evaluate the efficacy of frovatriptan when used at the early stage (International Headache Society [IHS] Grade 1) of MM compared with patients' current treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Had MM headaches occurring between Day -2 and Day +3 of menses
2. Had at least one year history of MM headaches
3. Had at least 8 MM headaches in the previous 12 menstrual cycles (1 year)
4. Had regular predictable menstrual periods (28 ± 4 days)

Exclusion Criteria:

1. Had a history of more than 15 headache days per month
2. As part of current MM treatment, used intermittent prevention with an analgesic (e.g., naproxen for 5 days to prevent the onset of MM)
3. Had a history of myocardial infarction, ischemic heart disease (or presented with symptoms or signs compatible with ischemic heart disease), coronary vasospasm (including Prinzmetal's variant angina), other significant underlying cardiovascular disease, or peripheral vascular disease
4. Had significant cerebrovascular disease, including basilar or hemiplegic migraine
5. Had uncontrolled hypertension: systolic blood pressure >180mmHg and diastolic blood pressure >95mmHg
6. Had severe hepatic or renal insufficiency
7. Used an analgesic medication (including both prescription and over-the-counter) for any reason >50% of days per month

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 192 (Actual)
Dates: Start 2005-09; Primary Completion 2006-02 (Actual); Study Completion 2006-02 (Actual)

PRIMARY OUTCOMES:
Headache pain severity | Visit - V1(Day 0), V2 (Day 28), V3 (Day 56)

SECONDARY OUTCOMES:
Occurrence and severity of MM symptoms associated with migraine headache pain (nausea, vomiting, photophobia, and phonophobia)
Occurrence and severity of functional impairment during menstrual migraine
Use of rescue medication and additional frovatriptan dose
Patient satisfaction with treatment
Patient preference of current vs. study treatment (end of study only)
Safety as assessed by occurrence of AEs

CONTACTS AND LOCATIONS:
Overall Officials: Sr. Director, Study Director — Endo Pharmaceuticals
Locations (21):
- United States (21):
  - Stratford, Connecticut
  - Clearwater, Florida
  - Jacksonville, Florida
  - Largo, Florida
  - Tampa, Florida
  - Blackwood, New Jersey
  - New York, New York
  - Plainview, New York
  - Vestal, New York
  - Burlington, North Carolina
  - Raleigh, North Carolina
  - Salisbury, North Carolina
  - Winston-Salem, North Carolina
  - Cincinnati, Ohio
  - West Chester, Ohio
  - Norristown, Pennsylvania
  - Philadelphia, Pennsylvania
  - Saint Petersburg, Pennsylvania
  - Upland, Pennsylvania
  - Nashville, Tennessee
  - Houston, Texas

REFERENCES:
- [Derived] MacGregor EA, Victor TW, Hu X, Xiang Q, Puenpatom RA, Chen W, Campbell JC. Characteristics of menstrual vs nonmenstrual migraine: a post hoc, within-woman analysis of the usual-care phase of a nonrandomized menstrual migraine clinical trial. Headache. 2010 Apr;50(4):528-38. doi: 10.1111/j.1526-4610.2010.01625.x. Epub 2010 Mar 2. PMID 20236340